CLINICAL TRIAL: NCT01060605
Title: Effects of Pre-transplant Rapamycin Treatment and Tacrolimus Levels on the Outcome of Islet Transplantation Alone in Patients Receiving Edmonton Protocol.
Brief Title: Pre Transplant Rapamycin Treatment in Islet Transplantation Alone
Acronym: ITA-Rp
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Ministry of Education, Universities and Research, Italy (Other); Juvenile Diabetes Research Foundation (Other); Telethon-JDRF Center for Beta cell replacement: clinical core. (Unknown)
Responsible Party: Antonio Secchi, IRCCS San Raffaele
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: emendament 2001 to C99B901251
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: islet transplantation; insulin independence; C-peptide secretion
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rapamycin pre transplant (Experimental): Pre-transplant rapamycin is administered for at least four weeks prior to the first islet infusion at the dose of 0.1 mg/kg (target trough levels: 8-10 ng/mL).
  Interventions: Drug: rapamycin

INTERVENTIONS:
Drug: rapamycin — Pre-transplant rapamycin is administered for at least four weeks prior to the first islet infusion at the dose of 0.1 mg/kg (target trough levels: 8-10 ng/mL).
  Other Names: Rapamune

SUMMARY:
Numerous changes to the original Edmonton protocol have been proposed in the attempt of improving the still unsatisfactory long-term function of ITA. Rapamycin may blunt the early inflammatory response to islet transplantation in the liver, thus favoring islet engraftment.

Aim of the investigators study was to evaluate the effect of a pre-transplant treatment with rapamycin in patients with type 1 diabetes receiving islet transplant alone and immunosuppression according to the Edmonton protocol.

DETAILED DESCRIPTION:
Pre-transplant rapamycin is administered for at least four weeks prior to the first islet infusion at the dose of 0.1 mg/kg (target trough levels: 8-10 ng/mL). During the pre-transplant rapamycin treatment rapamycin trough levels, renal and liver function, white blood cells count, total lymphocytes and lymphocytes subpopulations, hemoglobin, fibrinogen, cross-linked fibrin degradation products, C-reactive protein, exogenous insulin requirement every week for the first month, and monthly thereafter are measured. Induction and maintenance immunosuppressive regimen after each islet infusion is administered according to the Edmonton protocol (daclizumab, rapamycin, target trough levels: 12-15 ng/mL during the first 3 months and 10-12 ng/mL thereafter and tacrolimus 2 mg/day,target trough levels: 4-6 ng/mL). Islets are infused into the liver through the portal vein under local anesthesia Portography is performed before and after infusion. The islet function is evaluated measuring fasting C-pep, EIR, and HbA1c, immediately before the first islet infusion and subsequently every day for the first week, and then weekly for the first month ; every month after the last islet infusion for the first year and every 6 month thereafter.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes
* ≥5 years of type 1 diabetes
* hypoglycaemia unawareness
* progression of chronic complications of diabetes despite intensive insulin regimen

Exclusion Criteria:

* overt kidney disease
* chronic liver disease
* hepatic haemangioma
* severe cardiomyopathy
* untreated coronary artery disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2001-10; Primary Completion 2005-12 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Evidence of insulin independence with adequate control of blood glucose (<140 mg/mL fasting; < 180 mg/mL post prandial, after the final infusion | 1 year

SECONDARY OUTCOMES:
basal and stimulated C-peptide levels | weekly within 1st month; monthly for 1 year
glycated haemoglobin | monthly
rapamycin and tacrolimus trough levels | every week for the first month, and monthly thereafter
renal and liver function, white blood cells count, total lymphocytes and lymphocytes subpopulations (CD24, CD19), hemoglobin, fibrinogen (FG), cross-linked fibrin degradation products, C-reactive protein (CRP) | every week for the first month, and monthly thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Secchi, MD, Principal Investigator — Transplant Unit, IRCCS San Raffaele
Locations (1):
- Transplant Unit, IRCCS San Raffaele, Milan, Italy

REFERENCES:
- [Derived] Benedini S, Ermetici F, Briganti S, Codella R, Terruzzi I, Maffi P, Caldara R, Secchi A, Nano R, Piemonti L, Alejandro R, Ricordi C, Luzi L. Insulin-mimetic effects of short-term rapamycin in type 1 diabetic patients prior to islet transplantation. Acta Diabetol. 2018 Jul;55(7):715-722. doi: 10.1007/s00592-018-1141-z. Epub 2018 Apr 13. PMID 29654388
- [Derived] Piemonti L, Maffi P, Monti L, Lampasona V, Perseghin G, Magistretti P, Secchi A, Bonifacio E. Beta cell function during rapamycin monotherapy in long-term type 1 diabetes. Diabetologia. 2011 Feb;54(2):433-9. doi: 10.1007/s00125-010-1959-6. Epub 2010 Nov 3. PMID 21046356